CLINICAL TRIAL: NCT05343299
Title: Evaluation of Postoperative Experience of Two WALANT-type Modes of Anesthesia (Lidocaine Alone or Combined With Ropivacaine) Used in Ambulatory Surgery of the Upper Limb. A Single-center Prospective Randomized, Single-blind Study
Brief Title: Postoperative Experience of 2 WALANT-type Modes of Anesthesia Used in Ambulatory Surgery of the Upper Limb.
Acronym: ROPIWA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIMAO/2021-1/YG-01; 2021-006493-23 (EudraCT Number)
Record Dates: First submitted 2022-04-15; First posted 2022-04-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia, Local; Hand Surgery; Wrist Surgery; Elbow Surgery
Keywords: lidocaine,; ropivacaine,; carpal tunnel syndrome,; trigger finger
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder | interventions — Anesthesia, Local; Lidocaine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized, single-blind superiority study comparing two management modalities in WALANT-type anesthesia for ambulatory hand surgery: addition of ropivacaine to lidocaine (experimental group) versus lidocaine alone (control group).
  Jardé Law Research Involving Human Persons category 1
Who Masked: Participant, Investigator
Masking Description: The patient will be blinded to his or her anesthesia protocol. The investigating physician who performs the anesthesia and surgery will be different from the evaluators (IDE, hospital CRA, evaluating physician) who will be blinded to the patient's assignment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing hand surgery with a combination of lidocaine and ropivacaine (Experimental): Patients undergoing Wide Awake Local Anesthesia No Tourniquet -type hand surgery with lidocaine
  Interventions: Combination Product: Ambulatory surgery under a combination of Lidocaine and Ropivacaine
- Patients undergoing hand surgery with lidocaine alone (Active Comparator): Patients undergoing Wide Awake Local Anesthesia No Tourniquet -type hand surgery with lidocaine
  Interventions: Combination Product: Ambulatory surgery under Lidocaine alone

INTERVENTIONS:
Combination Product: Ambulatory surgery under Lidocaine alone — In this conventional procedure group, the anesthetic solution is administered subcutaneously and by infiltration into the surgical area. A maximum volume of 20 ml (dose dictated by the operation) of the solution is thus injected by the operator: Lidocaine 10mg/mL combined with adrenaline 0.005mg/mL administered at a dose of 10 to 20 mL, i.e. a total of 50 to 200 mg of lidocaine.
  Other Names: Local anesthesia with lidocaine alone
  Arms: Patients undergoing hand surgery with lidocaine alone
Combination Product: Ambulatory surgery under a combination of Lidocaine and Ropivacaine — In this experimental procedure group, the anesthetic solution is administered subcutaneously and by infiltration into the surgical area. A maximum volume of 20 ml (dose dictated by the operation) of the solution is thus injected by the operator: Lidocaine 10mg/mL combined with adrenaline 0.005mg/mL administered at a dose of 18 mL + ropivacaine 7.5 mg/mL 2 mL or 15 mg. For a total of 20 mL: lidocaine 9mg/mL, ropivacaine 0.75 mg/mL, adrenaline 0.005 mg/mL
  Other Names: Local anesthesia with lidocaine and ropivacaine
  Arms: Patients undergoing hand surgery with a combination of lidocaine and ropivacaine

SUMMARY:
Distal surgery of the upper limb under local anesthesia using the WALANT technique (Wide Awake Local Anesthesia No Tourniquet) has become the standard care in orthopedic surgery. The principle is that the operator infiltrates the whole surgical area with a 1% lidocaine solution combined with adrenaline (diluted to 1/200,000) so that all distal surgery of the upper limb can be performed without a tourniquet. Thus, the perioperative course and management of the patient in the operating room and the constraints inherent to general anesthesia are largely reduced. Also, the material cost is considerably reduced. However, WALANT often induces significant pain when the patient leaves the operating room to return home. This effect is related to the pharmacological formulation of lidocaine which has a short half-life (< 3h). To reduce this inconvenience of early block removal, adding a local anesthetic with a longer duration of action (ropivacaine) to lidocaine would extend the duration of the analgesic, improving postoperative experience and satisfaction. The main objective of this research is to evaluate the effect of two WALANT anesthesia protocols (with or without the addition of ropivacaine) on the postoperative experience of patients (QoR-40 questionnaire) 48 hours after outpatient hand surgery.

DETAILED DESCRIPTION:
Secondary objectives include the evaluation of short-term pain (Day 0 to Day 7), chronicisation of pain at 3 months, patient satisfaction regarding perioperative management and tolerance in both groups.

This is a monocentric, prospective, randomized, single-blind study. 80 adult patients, eligible for outpatient surgery under under WALANT for hand surgery such as carpal tunnel, stub finger, Dupuytren's disease or elbow surgery such as ulnar nerve compression and lacertus fibrosus syndrome, will be recruited during their care in the orthopedic and trauma surgery department at Nîmes University Hospital over an estimated period of 12 months. After receiving information, the intervention visit will be planned within 21 days. After collecting consent and checking the selection criteria, patients will be randomized (1:1 stratified according to hand/elbow surgery) for a procedure under WALANT anesthesia with 10 to 20 ml of 1% lidocaine (10 mg/mL) (depending on the procedure) combined with adrenaline (0.005mg/ml) with or without the addition of 15mg ropivacaine. An evaluation of the pain via a visual analog scale (0 to 10) will be carried out before discharge from the service and by telephone on Day 1 according to the current care then at Days 2 and 3 and 7 for the research. The patients will also have to answer questionnaires on their perioperative management (Evaluation of the experience of local anaesthesia or EVAN-LR) before leaving the department and then on the postoperative experience (Quality of Recovery or QoR-40) at D2 and the possible "chronicisation" of pain at 3 months (neuropathic pain or DN4) by telephone. Possible adverse events will be collected up to D7.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for outpatient surgery under WALANT for:
* Hand surgery such as carpal tunnel, stub finger, Dupuytren's disease;
* Elbow surgery such as ulnar nerve compression and lacertus fibrosus syndrome.
* Patient with free and informed consent.
* Patient with signed consent form.
* Patient affiliated to or beneficiary of a health insurance plan.

Exclusion Criteria:

* Ischemic vascular disorders such as severe Raynaud's disease, Buerger's disease, diabetic microangiopathy.
* Scleroderma.
* Known allergy to ropivacaine or lidocaine and possibility of cross-allergy with other amide-bound local cross-allergy with other local anesthetics with amide linkage.
* Severe hepatic impairment
* Acute porphyria.
* Intravascular anesthesia.
* Anesthesia by local infiltration in the extremities
* Coronary insufficiency.
* Ventricular rhythm disorders.
* Severe arterial hypertension.
* Obstructive cardiomyopathy.
* Hyperthyroidism.
* Hypovolemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Experimental group: experience of patients in the Lidocaine + Ropivacaine group | 48 hours after surgery
  The postoperative experience will be evaluated by the Quality of Recovery questionnaire (QoR-40) at 48 h postoperative.
  This questionnaire includes sections on comfort, pain, support, emotions and physical independence. Each section has questions to be answered on a scale of 1 to 5 in which 1 = very poor and 5 = excellent.
Control group: experience of patients in the Lidocaine alone group | 48 hours after surgery
  The postoperative experience will be evaluated by the Quality of Recovery questionnaire (QoR-40) at 48 h postoperative.
  This questionnaire includes sections on comfort, pain, support, emotions and physical independence. Each section has questions to be answered on a scale of 1 to 5 in which 1 = very poor and 5 = excellent.

SECONDARY OUTCOMES:
Pain on a numerical visual analog scale : Experimental group | Day 0
  Pain will be evaluated on a numerical visual analog scale in the experimental group.
  The scale ranges from 0 to 10 in which 0 = no pain and 10 = worst possible pain.
Pain on a numerical visual analog scale : Experimental group | Day 1
  Pain will be evaluated on a numerical visual analog scale in the experimental group.
  The scale ranges from 0 to 10 in which 0 = no pain and 10 = worst possible pain.
Pain on a numerical visual analog scale : Experimental group | Day 2
  Pain will be evaluated on a numerical visual analog scale in the experimental group.
  The scale ranges from 0 to 10 in which 0 = no pain and 10 = worst possible pain.
Pain on a numerical visual analog scale : Experimental group | Day 7
  Pain will be evaluated on a numerical visual analog scale in the experimental group.
  The scale ranges from 0 to 10 in which 0 = no pain and 10 = worst possible pain.
Neuropathic pain according to the DN4 questionnaire: Experimental group | At 3 months
  Pain in the experimental group will be evaluated by telephone using the DN4 questionnaire. This is a clinician-administered questionnaire consisting of 10 items. Seven items related to pain quality (i.e. sensory and pain descriptors) are based on an interview with the patient and 3 items based on the clinical examination. The DN4 (which stands for Douleur Neuropathique 4 i.e. Neuropathic Pain 4) is one of the questionnaires that can be useful in diagnosing neuropathic pain. It was initially written in French but immediately translated into English by the same team. The scale has been widely used since 2005 due to its simplicity. It evaluates neuropathic pain following central and peripheral neurological lesions. It is also used for diagnostic purposes, allowing the clinician to determine whether the pain is of neuropathic origin.This questionnaire has been well validated by a number of studies.
Satisfaction with perioperative management: Experimental group according to the EVAN-LR questionnaire | Day 0
  Patient satisfaction with perioperative management will be evaluated using the EVAN-LR (Evaluation du Vécu de l'Anesthésie LocoRégionale = Assessment of the Experience of Locoregional Anesthesia) self-reported questionnaire. This questionnaire, which specifically assesses the satisfaction of patients undergoing regional anesthesia, comprises 19 items, structured in a global index and five dimensions: Attention, Information, Discomfort, Waiting, and Pain. The consequences of staying alert during regional anesthesia are specifically addressed by two items.
Clinical or biological adverse events: Experimental group | From Day 0 to Day 2
  All clinical or biological adverse events will be recorded on the electronic reporting form from Day 0 up to Day 2. These include bleeding, hematoma, rehospitalization, paresthesia, nausea and vomiting after removal of anesthesia.
Pain on a visual numerical scale : Control group | Day 0
  Pain will be evaluated on a visual numerical scale in the control group
Pain on a visual numerical scale : Control group | Day 1
  Pain will be evaluated on a visual numerical scale in the control group
Pain on a visual numerical scale : Control group | Day 2
  Pain will be evaluated on a visual numerical scale in the control group
Pain on a visual numerical scale : Control group | Day 7
  Pain will be evaluated on a visual numerical scale in the control group
Neuropathic pain according to the DN4 questionnaire: Control group | At 3 months
  Pain in the control group will be evaluated by telephone using the DN4 questionnaire. This is a clinician-administered questionnaire consisting of 10 items. Seven items related to pain quality (i.e. sensory and pain descriptors) are based on an interview with the patient and 3 items based on the clinical examination. The DN4 (which stands for Douleur Neuropathique 4 i.e. Neuropathic Pain 4) is one of the questionnaires that can be useful in diagnosing neuropathic pain. It was initially written in French but immediately translated into English by the same team. The scale has been widely used since 2005 due to its simplicity. It evaluates neuropathic pain following central and peripheral neurological lesions. It is also used for diagnostic purposes, allowing the clinician to determine whether the pain is of neuropathic origin.This questionnaire has been well validated by a number of studies.
Satisfaction with perioperative management according to the EVAN-LR questionnaire Control group | Day 0
  Patient satisfaction with perioperative management will be evaluated using the EVAN-LR (Evaluation du Vécu de l'Anesthésie LocoRégionale = Assessment of the Experience of Locoregional Anesthesia) self-reported questionnaire. This questionnaire, which specifically assesses the satisfaction of patients undergoing regional anesthesia, comprises 19 items, structured in a global index and five dimensions: Attention, Information, Discomfort, Waiting, and Pain. The consequences of staying alert during regional anesthesia are specifically addressed by two items.
Clinical or biological adverse events: Control group | From Day 0 to Day 2
  All clinical or biological adverse events will be recorded on the electronic reporting form from Day 0 up to Day 2. These include bleeding, hematoma, rehospitalization, paresthesia, nausea and vomiting after removal of anesthesia.

OTHER OUTCOMES:
Sex of patients in the Experimental group | Day 0
  Male/Female
Age of patients in the Experimental group | Day 0
  In years
Weight of patients in the Experimental group | Day 0
  In kilograms
Height of patients in the Experimental group | Day 0
  In centimeters
Body Mass Index of patients in the Experimental group | Day 0
  BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Sex of patients in the Control group | Day 0
  Male/Female
Age of patients in the Control group | Day 0
  In years
Weight of patients in the Control group | Day 0
  In kilograms
Height of patients in the Control group | Day 0
  In centimeters
Body Mass Index of patients in the Control group | Day 0
  BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.

CONTACTS AND LOCATIONS:
Locations (1):
- Yann GRICOURT, Nîmes, Gard, France

REFERENCES:
- [Result] Gricourt Y, Occean BV, Favrelle A, Chevallier T, Mares O, Cuvillon P. Mixture of Lidocaine and Ropivacaine as a Local Anesthetic in WALANT Surgery: A Prospective Randomized Study. J Hand Surg Am. 2025 Jul;50(7):790-796. doi: 10.1016/j.jhsa.2025.03.010. Epub 2025 Apr 24. PMID 40272357